CLINICAL TRIAL: NCT07274904
Title: Evaluating Palliative Care Delivery: A Randomized Controlled Trial of Virtual Versus In-Person Approaches
Brief Title: Virtual Versus In-Person Approaches
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al Al Bayt University, Jordan (Other)
Collaborators: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Mohammad Al Qadire, Professor, Al Al Bayt University, Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-2024/25
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Palliative Care, Patient Care
Keywords: Palliative care; Virtual; Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telepalliative Care (Experimental): Participants assigned to this arm will receive early palliative care delivered primarily through scheduled virtual visits. Consultations will occur approximately every four weeks using secure video-conferencing platforms or, when necessary, telephone calls. A multidisciplinary palliative care team-including physicians, nurses, and other supportive care providers-will conduct symptom assessments, provide management recommendations, offer psychosocial support, and engage in care planning. Caregivers may join the virtual sessions when available. Additional follow-up contacts may be arranged to address urgent concerns or symptom changes. The clinical content is equivalent to standard in-person palliative care; only the delivery modality differs.
  Interventions: Other: Virtual Early Palliative Care
- In-Person Palliative Care (Active Comparator): Participants assigned to the control arm will receive standard early palliative care through face-to-face clinic visits at the King Hussein Cancer Center every four weeks. Care is provided by a multidisciplinary team consisting of physicians, nurses, social workers, and other supportive care professionals. Services include routine symptom monitoring, adjustment of treatment plans, psychosocial support, and additional assessments as clinically indicated. All clinical content follows evidence-based palliative care guidelines. The primary difference from the intervention arm is that care is delivered in person rather than virtually.
  Interventions: Other: Standard In-Person Early Palliative Care

INTERVENTIONS:
Other: Virtual Early Palliative Care — This intervention consists of structured early palliative care delivered primarily through secure video-based consultations approximately every four weeks. Sessions are conducted by a multidisciplinary palliative care team and include symptom assessment, management recommendations, psychosocial support, and care planning. Telephone calls may be used when video is not feasible. The clinical content mirrors standard palliative care, but all routine visits are conducted remotely rather than in person.
  Arms: Telepalliative Care
Other: Standard In-Person Early Palliative Care — This intervention involves face-to-face early palliative care visits conducted on-site at the King Hussein Cancer Center every four weeks. Care is provided by a multidisciplinary team and includes routine symptom evaluation, treatment adjustments, psychosocial support, and additional assessments as needed. The clinical services follow standard palliative care guidelines. This arm differs from the intervention arm only in delivery mode, as all visits occur in person.
  Arms: In-Person Palliative Care

SUMMARY:
This randomized controlled trial evaluates the effectiveness of two models of early palliative care delivery for adults with cancer: virtual care provided through scheduled video consultations and standard in-person clinic visits. Early palliative care aims to improve quality of life, manage symptoms, and support patients and families throughout the course of serious illness. Although in-person services are well established, access barriers may limit their use, and virtual care may offer a feasible alternative.

Participants are randomly assigned to receive either virtual early palliative care or in-person early palliative care. Both models include structured assessments of physical and psychological symptoms, communication and decision-making support, and routine follow-up with a palliative care specialist. Outcomes are assessed at baseline and at 3, 6, and 12 months. Primary and secondary outcomes include quality of life, symptom burden, psychological distress, patient satisfaction, and healthcare utilization.

The purpose of the study is to determine whether virtual early palliative care delivers outcomes comparable to those of traditional in-person care. The results may inform future models of palliative care delivery by identifying approaches that improve accessibility while maintaining high-quality patient support.

DETAILED DESCRIPTION:
Evaluating Palliative Care Delivery: A Randomized Controlled Trial of Virtual Versus In-Person Approaches Background Palliative care is a patient- and family-centered approach that seeks to improve quality of life and alleviate suffering among individuals with serious or life-threatening illness (Wantonoro et al., 2022). It emphasizes relief from pain and other distressing symptoms while addressing psychosocial, emotional, and spiritual concerns (World Health, 2018). Unlike traditional perceptions of palliative care as end-of-life treatment, contemporary definitions underscore its integration early in the disease trajectory, delivered concurrently with curative or life-prolonging therapies (Wantonoro et al., 2022). This shift toward early integration recognizes that patients often experience significant symptom burden and psychosocial distress from the point of diagnosis of advanced illness, and that timely intervention can mitigate these challenges while fostering better coping and decision-making.

Historically, palliative care has been delivered predominantly in person through hospital-based services, outpatient clinics, or home-based programs (Ferrell et al., 2017). These models often involve interdisciplinary teams of physicians, nurses, social workers, and spiritual care providers who collaborate to provide holistic care (Ferrell et al., 2017). While effective, such models are resource intensive and may be geographically limited, especially in regions with sparse specialist availability. Technological advances and the COVID-19 pandemic accelerated the adoption of virtual modalities, demonstrating their potential to maintain continuity of care while reducing exposure risks and travel burdens (Calton et al., 2020).

Telepalliative care, including video consultations, telephone follow-ups, and digital platforms, has emerged as a feasible and effective alternative to in-person encounters. For instance, video consultations delivered by nurses in home-based settings have been shown to be feasible and cost-effective with strong patient and family engagement (Ma et al., 2025). Culturally tailored video consultations have been successfully implemented in rural hospitals lacking palliative services (Bakitas et al., 2025). Early palliative care via video visits has demonstrated equivalent outcomes to in-person care. Moreover, patients and families report that telepalliative care improves access, convenience, and satisfaction, particularly when integrated with standard care workflows (Greer et al., 2024; Mathews et al., 2023). Telehealth models are particularly appealing in contexts where specialist shortages and geographic inequities limit access.

With the growing adoption of telemedicine, attention has turned to whether virtual palliative care can achieve outcomes comparable to traditional in-person delivery (Greer et al., 2024; Sebastian et al., 2024; Yang et al., 2024). A recent systematic review and meta-analysis of randomized controlled trials in patients with chronic heart failure evaluated integrated palliative care delivered through telehealth (Sebastian et al., 2024). They found significant improvements in quality of life-measured by the Kansas City Cardiomyopathy Questionnaire and the Functional Assessment of Chronic Illness Therapy-Palliative Care scale-as well as reduced hospitalizations when compared to usual care (Sebastian et al., 2024). Similarly, a systematic review and meta-analysis focusing on informal caregivers of palliative care patients was condcuted (Yang et al., 2024). Their analysis showed that telemedicine interventions influenced caregiver outcomes, including burden, anxiety, depression, and quality of life, underscoring the broader impact of virtual models on families (Yang et al., 2024).

In addition to meta-analyses, recent large randomized controlled trials have provided high-quality evidence. A multisite randomized clinical trial involving 1,250 patients with advanced non-small cell lung cancer was condcuted (Greer et al., 2024). Participants were randomized to receive early palliative care either through secure video visits or through in-person sessions across 22 United States cancer centers. At 24 weeks, quality of life outcomes-assessed with the Functional Assessment of Cancer Therapy-Lung scale-were statistically equivalent between groups. There were also no significant differences in mood, coping, satisfaction, or health care utilization. However, caregiver participation was modestly lower in the telehealth arm, highlighting the need for tailored strategies to optimize family engagement in virtual settings (Greer et al., 2024).

Collectively, these findings provide compelling evidence that telepalliative care can deliver outcomes comparable to traditional models, while also identifying important considerations for caregiver involvement. Despite these advances, the majority of palliative care research has been conducted in high-income countries (HICs). Globally, an estimated 40 million people require palliative care annually, yet only 14% receive it, with the vast majority of unmet need concentrated in low- and middle-income countries (LMICs) (World Health Organization, 2020). Barriers in LMICs include limited specialist workforce, geographic inaccessibility, weak health system infrastructure, and competing healthcare priorities (Clark et al., 2018). Even where palliative care services exist, access is frequently inequitable, favoring urban centers and wealthier populations.

Palliative care is widely recognized as an essential component of comprehensive cancer care, yet global inequities in access remain stark. Telepalliative care has emerged as a promising strategy to extend specialist services, reduce travel burdens, and facilitate scalable models of early intervention, particularly where workforce shortages and geographic barriers limit access. Despite these advantages, robust comparative data evaluating the effectiveness of telepalliative care versus in-person delivery are lacking in LMICs. Evidence HICs may not be directly generalizable due to fundamental differences in infrastructure, digital literacy, cultural norms, and health system capacity. Recent systematic reviews reinforce this evidence gap. A comprehensive review of telehealth interventions in oncology concluded that while telepalliative care can improve psychological outcomes and enhance access, reporting on physical symptom burden and other core aspects of patient well-being remains inconsistent (Mathews et al., 2023). This highlights the need for research that rigorously evaluates the impact of telepalliative models on the physical dimensions of suffering, including pain, fatigue, and other distressing symptoms. Importantly, the Oncology Nursing Society's (ONS) current research agenda explicitly identifies precision symptom science and integration of palliative care into routine oncology practice as critical research priorities, underscoring the urgency of addressing gaps in symptom-focused evidence (Rosenzweig et al., 2024).

Taken together, these gaps establish a compelling rationale for the proposed study. By generating locally relevant, high-quality evidence on telepalliative care in LMICs, the research will address both the scientific need for data on physical symptom burden and the strategic research priorities articulated by international professional bodies. The findings will provide critical guidance for policymakers, health systems, and clinicians on how best to integrate telepalliative care into diverse contexts, ensuring that limited resources are leveraged effectively to improve patient and caregiver outcomes. Therefor, the purpose of this study is to evaluate the effectiveness, feasibility, and acceptability of tele palliative care among cancer patients in Jordan. Specifically, the study aims to determine whether tele palliative care can provide outcomes comparable to in-person care in terms of quality of life, symptom burden, and healthcare facility utilization.

Objectives and Hypotheses Primary Objectives

1. To evaluate whether telepalliative care provides quality of life outcomes comparable to in-person palliative care among cancer patients in Jordan.
2. To assess whether telepalliative care results in a comparable level of symptom burden relative to in-person palliative care.
3. To determine whether patient satisfaction with care in the telepalliative model is comparable to satisfaction reported in in-person care.

Null Hypothesis: Among cancer patients in Jordan, there are no significant differences between telepalliative care and in-person care with respect to quality of life, symptom burden, and satisfaction with care.

Secondary Objectives

1. To evaluate the effect of telepalliative care on psychological distress compared to in-person care.
2. To compare the rates of unplanned hospital visits between patients receiving telepalliative versus in-person palliative care.
3. To compare hospital admissions and length of stay between the two models of care.

Null Hypothesis: Telepalliative care does not differ significantly from in-person palliative care in terms of psychological distress, frequency of unplanned hospital visits, number of admissions, and length of hospital stay.

Methods Design This study will be conducted as a single-site, non-blinded randomized clinical trial, in which eligible participants will be randomly assigned to receive either telepalliative care or standard in-person palliative care. The non-blinded design is appropriate given the nature of the intervention, as masking participants and providers to the mode of care delivery is not feasible.

Setting The study will be conducted at the King Hussein Cancer Center (KHCC) in Amman, Jordan. KHCC is a major referral center for cancer care in the country and provides a range of oncology and supportive care services. Its palliative care program includes inpatient and outpatient services, consultation support, and a home care component delivered by an interdisciplinary team of physicians, nurses, social workers, psychologists, and spiritual care providers. The center also offers a fellowship in hospice and palliative medicine accredited by the Jordanian and Arab Medical Councils. This setting provides access to a diverse patient population and an established palliative care infrastructure in which to evaluate telepalliative care interventions.

Sample The sample will include patients referred to palliative care services within the KHCC. Participants will be eligible for inclusion if they are adults aged 18 years or older, diagnosed with solid tumours at any stage, referred to palliative care services at the KHCC, able to read and write in Arabic, and capable of providing informed consent. Patients will be excluded if they have severe cognitive impairment or psychiatric conditions that limit their ability to consent or participate meaningfully, are critically ill or receive end-of-life care where participation would cause an undue burden or are unable to participate in telehealth interventions due to lack of access to the necessary technology and absence of caregiver support.

Sampling size The sample size calculation was based on the planned statistical analysis. An independent t-test will be used to compare outcomes between the control and intervention arms of the study. Using G*Power version 3.1, and assuming a two-tailed test with a significance level of α = 0.05, a medium effect size (Cohen's d = 0.5), power = 0.95, and a 1:1 allocation ratio, the required sample size was estimated at 105 participants per group. To account for an anticipated attrition rate of 20%, the final target sample size will be 252 participants, with 126 allocated to each group.

Study Arms The intervention Arm (Telepalliative Care) Participants randomised to the telepalliative care arm will receive scheduled palliative care consultations every four weeks, delivered primarily through virtual modalities. Visits will be conducted using secure video-conferencing platforms or, when necessary, telephone calls. The clinical team will include physicians, nurses, and other palliative care professionals, who will provide symptom assessment, management recommendations, psychosocial support, and care planning. Caregivers will be encouraged to join virtual sessions when available. Additional follow-up contacts may be arranged as needed to address emerging concerns, medication adjustments, or urgent symptom management.

Control Arm (In-Person Palliative Care) Participants randomised to the in-person care arm will receive standard palliative care services through face-to-face appointments at the King Hussein Cancer Center every four weeks. Care will be delivered by a multidisciplinary palliative care team, including physicians, nurses, social workers, and other supportive care providers. Services will include routine symptom monitoring, adjustment of treatment plans, and supportive counselling. Unplanned visits or additional assessments will be scheduled as clinically indicated.

Both arms will follow evidence-based palliative care guidelines and will have access to the same range of clinical expertise. The primary difference between the two arms will be the mode of service delivery (virtual versus in-person).

Randomaiztion All patients who are referred to the palliative care services will be invited to participate during their routine clinic visit. After confirming eligibility and obtaining informed consent, participants will be randomized in a 1:1 ratio to either the telepalliative care group or the in-person palliative care group. Randomization will be conducted using a computer-generated random allocation sequence to ensure balance between groups and to minimize selection bias. The allocation sequence will be concealed in sealed, opaque envelopes that will be opened sequentially after enrollment.

Outcomes Measurements Quality of Life (EORTC QLQ-C15-PAL) Quality of life will be assessed using the EORTC QLQ-C15-PAL, a 15-item short form of the QLQ-C30 developed for use in palliative cancer care (Groenvold et al., 2006). The instrument includes two multi-item functional scales (physical functioning: 3 items; emotional functioning: 2 items), two multi-item symptom scales (fatigue: 2 items; pain: 2 items), five single-item symptom measures (dyspnea, insomnia, nausea/vomiting, appetite loss, constipation), and one global health status/quality-of-life item. Most items are rated on a 4-point Likert scale from "not at all" to "very much," and the global QoL item uses a 7-point scale. Scores will be transformed to a 0-100 scale, where higher scores represent better functioning or greater symptom burden, depending on the domain. An Arabic version has been validated in Jordanian patients with advanced cancer, showing satisfactory reliability with Cronbach's alpha values = .898 (Alawneh et al., 2016).

Symptom Burden (MD Anderson Symptom Inventory, MDASI) Symptom burden will be measured using the MD Anderson Symptom Inventory (MDASI), developed to assess the severity of multiple cancer-related symptoms and their interference with daily life (Cleeland et al., 2000). The tool consists of 19 items: 13 assess symptom severity (e.g., pain, fatigue, nausea, disturbed sleep, shortness of breath) and 6 assess interference with functioning (e.g., general activity, mood, work, enjoyment of life, relations with others, walking). Each item is scored on a 0-10 numeric scale, with higher scores indicating greater severity or interference. Arabic versions have been validated in oncology populations, reporting Cronbach's alpha coefficients between 0.78 and 0.85, indicating strong internal consistency (Nejmi et al., 2010).

Patient Satisfaction (EORTC IN-PATSAT32) Patient satisfaction will be measured using the EORTC IN-PATSAT32, developed to assess satisfaction with doctors, nurses, and aspects of care organization in oncology (Bredart et al., 2005). The 32 items are grouped into subscales that evaluate communication, technical competence, interpersonal skills, availability, and organizational factors. Items are rated on 5-point Likert scales and transformed to 0-100 scores, with higher scores indicating greater satisfaction. The Arabic version demonstrated acceptable psychometric properties, with Cronbach's alpha values ranging from 0.72 to 0.95 across subscales, confirming its reliability in Arabic-speaking cancer populations (Obtel et al., 2017).

Psychological Distress (Hospital Anxiety and Depression Scale, HADS) Anxiety and depression will be measured with the Hospital Anxiety and Depression Scale (HADS), developed to detect these conditions in patients with physical illness while minimizing confounding by somatic symptoms (Zigmond & Snaith, 1983). The HADS includes 14 items, with 7 assessing anxiety (HADS-A) and 7 assessing depression (HADS-D). Each item is scored from 0 to 3, producing subscale scores ranging from 0 to 21. Standard cutoffs will be applied: 0-7 (normal), 8-10 (borderline), and ≥11 (probable case)(Zigmond & Snaith, 1983). The Arabic version has been validated in cancer patients, showing excellent reliability (Cronbach's α = 0.83 for anxiety, 0.77 for depression) (Terkawi et al., 2017).

Sociodemographic Data, Patient clinical characteristics: Tumor type, cancer stage, date of diagnosis, performance status, etc. per electronic health record review. Patient health care utilization: PC visits, chemotherapy and radiation administration, emergency department visits, ICU admissions, hospitalizations, and location of death per electronic health record.

Sociodemographic and Clinical Characteristics. Sociodemographic data will be collected, including age, sex, marital status, education level, employment status, health insurance coverage, household income, and place of residence (urban versus rural). Clinical characteristics will be obtained from electronic health records and will include tumor type, cancer stage at diagnosis, date of diagnosis, prior treatments (surgery, chemotherapy, radiotherapy), and current treatment status.

Health Care Utilization Information on health service utilization will also be extracted from electronic health records. This will include the number of unplanned palliative care visits, chemotherapy and radiotherapy sessions, emergency department visits, intensive care unit admissions, and hospitalizations (including length of stay). These data will help assess the impact of telepalliative versus in-person care on healthcare resource use.

Data Collection procedure Data collection will commence only after obtaining ethical approval from the Institutional Review Boards of the university affiliated with the principal investigator and the King Hussein Cancer Center. At the initial clinic visit, all eligible patients will be screened, informed of the study, and invited to provide written informed consent. Baseline data will then be collected for both groups during this first face-to-face encounter. Sociodemographic and clinical information will be obtained through a secure online platform, and participants will complete baseline questionnaires measuring their quality of life, symptom burden, satisfaction with care, and psychological distress. Clinical information will also be extracted from the electronic health records.

Following the baseline assessment, participants will be randomised into either the telepalliative care arm or the in-person palliative care arm. In both groups, palliative care appointments will be scheduled every four weeks. If an appointment is missed, the research coordinator will contact the participant within 48 h of rescheduling, and the visit will be conducted within one week using the assigned mode of delivery.

Outcome data will be collected at baseline and at 3, 6, and 12 months using the same validated questionnaires. Healthcare utilisation outcomes, including unplanned palliative care visits, chemotherapy and radiotherapy sessions, emergency department visits, intensive care unit admissions, and hospitalisations (including length of stay), will be extracted from the electronic health records at the same intervals. To ensure data quality, entries were checked for completeness and accuracy, and discrepancies were verified against the source documents. All data will be de-identified, stored on password-protected servers, and made accessible only to the research team.

Ethical Considerations This study will be conducted in accordance with the principles outlined in the Declaration of Helsinki and its amendments. Ethical approval will be obtained from the Institutional Review Board (IRB) of the university affiliated with the principal investigator, followed by approval from the Institutional Review Board of the KHCC, prior to study initiation.

Participation will be voluntary. Patients will be provided with detailed verbal and written information about the study objectives, procedures, potential risks, and expected benefits in Arabic language. Informed consent will be obtained before enrolment, and participants will be assured that their refusal to participate or withdrawal from the study at any stage will not affect the quality of care they receive. Confidentiality will be strictly maintained. Each participant will be assigned a unique study identification number, and all data will be stored securely in password-protected electronic files that are accessible only to the research team. Identifiable personal information will not included in the publications or presentations of this study.

Given the nature of the study population, special attention will be paid to minimizing burden. The study interventions, telepalliative care and in-person palliative care, represent variations in standard clinical practice, and no participant will be deprived of essential care. If a participant experiences worsening symptoms or distress, appropriate clinical support will be provided immediately.

Data analysis Data will be analyzed using IBM SPSS Statistics version 30 (IBM Corp., Armonk, NY). Descriptive statistics will summarize baseline demographic and clinical characteristics. For the primary and secondary outcomes, independent t-tests will be used to compare mean scores between the intervention and control groups, and repeated-measures ANOVA will be applied to examine changes over time. All analyses will be conducted according to the intention-to-treat principle, with statistical significance set at α = 0.05 (two-tailed).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Diagnosed with a solid tumor at any stage
* Referred to palliative care services at the King Hussein Cancer Center (KHCC)
* Able to read and write in Arabic
* Capable of providing informed consent

Exclusion Criteria:

* Severe cognitive impairment that limits ability to consent or meaningfully participate
* Psychiatric conditions that interfere with ability to consent or participate
* Critically ill or receiving end-of-life care where participation would cause undue burden
* Inability to participate in telehealth interventions due to lack of access to necessary technology
* Absence of caregiver support when needed for telehealth participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Quality of life (EORTC QLQ-C15-PAL) | Baseline, 3 months, 6 months, and 12 months after randomization.
  Quality of life will be measured using the EORTC QLQ-C15-PAL, a 15-item questionnaire developed for palliative cancer care. It includes functional and symptom scales and a global quality-of-life item. Scores are transformed to a 0-100 scale, with higher scores indicating better functioning or greater symptom burden depending on the domain. Mean scores will be compared between telepalliative and in-person arms over time.
Symptom Burden (MD Anderson Symptom Inventory - MDASI) | Baseline, 3 months, 6 months, and 12 months after randomization.
  Symptom burden will be assessed using the MD Anderson Symptom Inventory (MDASI), a validated 19-item instrument that evaluates the severity of common cancer-related symptoms and the extent to which these symptoms interfere with daily functioning. Thirteen items measure symptom severity (e.g., pain, fatigue, disturbed sleep), and six items measure interference with activities, mood, and quality of life. Each item is scored on a 0-10 numeric scale, with higher scores indicating greater severity or interference. Mean symptom burden scores will be compared between telepalliative and in-person care groups over time.

SECONDARY OUTCOMES:
Patient Satisfaction (EORTC IN-PATSAT32) | Baseline, 3 months, 6 months, and 12 months after randomization.
  Patient satisfaction with palliative care services will be assessed using the EORTC IN-PATSAT32, a validated 32-item questionnaire measuring patients' perceptions of quality of care and quality of service provided by healthcare professionals. The instrument covers domains such as communication, interpersonal skills, information provision, technical skills, and organizational aspects of care. Scores are transformed to a 0-100 scale, with higher scores indicating greater satisfaction. Satisfaction levels will be compared between the telepalliative care and in-person care groups.

IPD SHARING:
Plan to Share IPD: No
The dataset includes sensitive clinical information from patients receiving palliative care, and the study team cannot ensure full de-identification without risk of re-identification due to the small population and the detailed nature of the clinical data. Ethical and regulatory requirements, including institutional policies and participant privacy protections, restrict the sharing of raw participant-level data. Aggregate results will be shared through publications and presentations.